CLINICAL TRIAL: NCT05739253
Title: Changes of Ascending Aortic Diameter in Patients Undergoing Transcatheter Aortic Valve Replacement
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-1602
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Aortic Stenosis; Ascending Aortic Dilatation; Bicuspid Aortic Valve
Keywords: Transcatheter aortic valve replacement; Ascending aortic diameter; Ascending aortic dilatation; Bicuspid aortic valve
MeSH Terms: conditions — Aortic Valve Stenosis; Bicuspid Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transfemoral TAVR for AS: Patients undergoing transfemoral transcatheter aortic valve replacement for aortic stenosis
  Interventions: Procedure: Transcatheter aortic valve replacement

INTERVENTIONS:
Procedure: Transcatheter aortic valve replacement — All patients undergo transfemoral transcatheter aortic valve replacement for aortic stenosis

SUMMARY:
The goal of this observational study is to assess the changes of ascending aortic diameter in patients undergoing transcatheter aortic valve replacement. The main questions it aims to answer are:

1. whether the ascending aortic diameter increases or remains stable after transcatheter aortic valve replacement, especially in patients with preoperative ascending aortic dilatation;
2. the determinants of postoperative ascending aortic dilatation.

DETAILED DESCRIPTION:
Ascending aortic (AA) dilatation occurs frequently in patients with aortic stenosis (AS). For patients who are candidates for transcatheter aortic valve replacement (TAVR), simultaneous repair of a dilatated AA is technically difficult. As the indications for TAVR have extended to low-risk patients and patients with bicuspid aortic valve , AA dilatation should be considered as a new criterion to refine risk stratification in patients undergoing TAVR. In this observational study, we aim to evaluate the changes of AA diameters and identify the determinants post-TAVR AA dilatation.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis defined as an aortic valve area of 1cm2 or less or an indexed aortic valve area of 0.6cm2/m2 or less;
* Presence of clinical symptoms defined as a New York Heart Association functional class of 2 or more;
* High risk of surgical aortic valve replacement;
* Suitability for a transfemoral vascular access.

Exclusion Criteria:

* Dominant aortic regurgitation;
* History of surgical or transcatheter aortic valve replacement;
* History of aortic surgery;
* Connective tissue disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The indication to perform transcatheter aortic valve replacement was based on a consensus by the Institutional Heart Team.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-03-21 (Estimated); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
Rate of ascending aortic dilatation | 1-year and 2-year
  The change of AA diameters (before the procedure and at the latest follow-up) divided by the follow-up period.

SECONDARY OUTCOMES:
Rate of all-cause mortality | 1-year and 2-year
  All-cause mortality during the follow-up period
Rate of adverse aortic events | 1-year and 2-year
  Aortic dissection, aortic rupture, and sudden death not attributable to other causes.

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Cardiovascular Disease, China & Fuwai Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] An K, Zhang F, Ouyang W, Pan X. Blood flow dynamics in the ascending aorta of patients with bicuspid aortic valve before and after transcatheter aortic valve replacement: a computational fluid dynamics study. BMC Cardiovasc Disord. 2024 Dec 20;24(1):717. doi: 10.1186/s12872-024-04394-w. PMID 39702010